CLINICAL TRIAL: NCT03922100
Title: A Phase I/II Study of NMS-03592088, a FLT3, KIT and CSF1R Inhibitor, in Patients With Relapsed or Refractory AML or CMML
Brief Title: Study of NMS-03592088 in Patients With Relapsed or Refractory AML or CMML
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped due to strategic reasons. The decision is not based on specific safety findings as the safety observed in the phase II part of the study is in line with what was reported in the phase I part.
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MKIA-088-001; 2018-002793-47 (EudraCT Number)
Record Dates: First submitted 2019-04-04; First posted 2019-04-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia (AML); Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Intervention Model Description: This is an open-label Phase I/II, first-in-human (FIH), non-randomized, multi-center study conducted in two parts: a Phase I including patients with AML and CMML and a Phase II exploratory study comprising two parallel cohorts of AML FLT3 mutated patients.
  The Phase II portion of the study is currently being conducted in EU only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMS-03592088 (Experimental): Phase I Dose Escalation
  * Schedule A - Starting dose of 20 mg/day
  * Schedule B - Starting dose of 120 mg/day
  Only one dose level open for enrollment except EU backfill cohorts.
  Phase II Dose Expansion (Exploratory) - (EU)
  Recommended Phase II Dose (RP2D) of NMS-03592088 in Phase 1
  * Cohort 1: Patients who have failed standard of care including venetoclax and gilteritinib based therapies
  * Cohort 2: Patients who have failed standard of care
  Interventions: Drug: NMS-03592088

INTERVENTIONS:
Drug: NMS-03592088 — Route of administration: Oral

SUMMARY:
The purpose of this study is to explore safety, tolerability, including the maximum tolerated dose and the recommended Phase II dose (RP2D), and antitumor activity of NMS-03592088 in adult patients with relapsed or refractory Acute Myeloid Leukemia (AML) or Chronic Myelomonocytic Leukemia (CMML).

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory disease who have failed standard therapy or are unsuitable for standard treatment, with one the following confirmed diagnosis: AML as defined by the European LeukemiaNet (ELN)
* Patients with confirmed diagnosis of AML as defined by the 2022 ELN recommendations
* Patients must have failed standard of care.
* Adult (age ≥ 18 years) patients
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* The interval from prior antitumor treatment to time of NMS-03592088 administration should be at least 2 weeks for any agents other than hydroxyurea.
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to NCI CTCAE version 5.0 Grade ≤1
* Adequate hepatic and renal function
* Patients must use highly effective contraception.
* Signed and dated IEC or IRB-approved informed consent form.

Exclusion Criteria:

* Current enrollment in another interventional clinical study
* Diagnosis of acute promyelocytic leukemia or Breakpoint cluster region-Abelson (BCR-ABL)-positive leukaemia
* Currently active second malignancy, except for adequately treated basal or squamous cell skin cancer and/or cone biopsied in situ carcinoma of the cervix uteri and/or superficial bladder cancer.
* Patients with known leukemia involvement of central nervous system (CNS)
* Hematopoietic stem cell transplantation (HSCT) within 3 months of treatment start and/or persistent non-hematologic toxicities of Grade ≥2 related to the transplant
* Active acute or chronic graft versus host disease (GVHD) requiring immunosuppressive treatment
* Patients with QTcF interval ≥ 480 milliseconds or with risk factors for torsade de pointes
* Pregnancy.
* Breast-feeding or planning to breast feed during the study or within 3 months after study treatment.
* Any of the following in the previous 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
* Known active, life threatening or clinically significant uncontrolled systemic infection.
* Known active gastrointestinal disease
* Known active gastrointestinal ulcer
* Other severe or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation.
* Known diagnosis of myasthenia gravis

US only:

* Signs or symptoms of myasthenia gravis or stroke during screening
* Patients with myasthenia gravis specific autoantibodies or any known history of myasthenia gravis (MG) autoantibodies at screening window
* Concomitant medications with the potential to cause de novo myasthenia gravis, worsening of myasthenia gravis or cause myasthenia gravis-like symptoms
* Uncontrolled hypertension, atrial fibrillation or flutter, ventricular arrhythmia or receiving treatment for cardiac rhythm disorder or diabetes that is not adequately controlled

Other protocol specific inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Phase I - Number of Participants with drug related first-cycle dose limiting toxicities (DLTs) | From the date of treatment initiation up to end of Cycle 1 (each Cycle is 28 days)
  DLTs will be classified according to NCI CTCAE version 5.0.
Phase II FLT3-ITD mut AML: Composite Complete Remission (CRc) Rate | From the date of treatment initiation up to end of study (approximately 1.5 years)
  Defined by the 2022 European LeukemiaNet (ELN) recommendations.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From the Informed Consent signature to 28 days after the last on-study treatment administration.
  Safety will be assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.).
Maximum plasma concentration (Cmax) of NMS-03592088 and its metabolites NMS-03593860 and NMS-03603422: | Phase 1 Dose Escalation and Dose Expansion Schedule A: Cycle 1 and Cycle 2 various timepoints; Phase 1 Dose Escalation Schedule B: Cycle 1, 2 and 3 various timepoints; Phase 1 Backfill Cycle 1 and Cycle 2 various timepoints (Each Cycle is 28 days)
  Plasma samples will be collected and used for pharmacokinetics assessments.
Time to maximum plasma concentration (Tmax) of NMS-03592088 and its metabolites NMS-03593860 and NMS-03603422: | Phase 1 Dose Escalation and Dose Expansion Schedule A: Cycle 1 and Cycle 2 various timepoints; Phase 1 Dose Escalation Schedule B: Cycle 1, 2 and 3 various timepoints; Phase 1 Backfill Cycle 1 and Cycle 2 various timepoints (Each Cycle is 28 days)
  Plasma samples will be collected and used for pharmacokinetics assessments.
Area under the plasma concentration versus time curve (AUC)] of NMS-03592088 and its metabolites NMS-03593860 and NMS-03603422: area under the plasma concentration versus time curve (AUC)] | Phase 1 Dose Escalation and Dose Expansion Schedule A: Cycle 1 and Cycle 2 various timepoints; Phase 1 Dose Escalation Schedule B: Cycle 1, 2 and 3 various timepoints; Phase 1 Backfill Cycle 1 and Cycle 2 various timepoints (Each Cycle is 28 days)
  Plasma samples will be collected and used for pharmacokinetics assessments.
Renal clearance of NMS-03592088 and its metabolites NMS-03593860 and NMS-03603422 excreted in urine (only Phase I) | Timepoints up to 24-hours post dose
Fraction of NMS-03592088 and its metabolites NMS-03593860 and NMS-03603422 excreted in urine (only Phase I) | Timepoints up to 24-hours post dose
Best response rate for participants with AML | From the date of treatment initiation up to end of study (approximately 1.5 years)
  Number and percentage of participants with CR, CRi, CRh, PR, MLFS, SD, No Response and Progressive Disease (PD).
Best response rate for participants with CMML | From the date of treatment initiation up to end of study (approximately 1.5 years)
  Number and percentage of participants with CR, CCR, PR, MR, CB and PD.
Overall Survival (OS) | From the date of treatment initiation until death or up to 1.5 years from patient's first dose, whichever comes first
  OS is defined as the time from the date of the first dose of study drug until the date of death for any cause.
Time to Response (TTR) | From the date of treatment initiation up to end of study (approximately 1.5 years)
  TTR is defined as the time from the first dose of study drug until the date of first response (CRc or PR).
Duration of Response (DoR) | From the date of first response up to end of study (approximately 1.5 years)
  Duration of response was defined as the time from the date of either first CRc or PR until the date of documented relapse of any type for participants who achieved CRc or PR.
Event-Free Survival (EFS) | From the date of treatment initiation until death or up to 1.5 years from patient's first dose, whichever comes first
  For patients with diagnosis of AML the primary analysis measures the time from the date of treatment initiation to the date of first documentation of disease progression or hematologic relapse after CR/CRh/CRi, treatment failure or death from any cause, whichever comes first.
  For patients with CMML, EFS will be defined as the time from treatment start until disease progression, relapse after CR, CCR, PR, MR or CB, treatment failure, or death from any cause, whichever comes first.
Relapse-free Survival (RFS) | From the date of treatment initiation until death or up to 1.5 years from patient's first dose, whichever comes first
  For patients with diagnosis of AML in the primary analysis it is measured only for patients achieving CR or CRi, and it is defined as the time from the date of first achievement of a CR/CRi until the date of relapse or death from any cause.
  For patients with CMML diagnosis, RFS will be measured from the date of first achievement of CR, CCR, PR, MR or CB until the date of relapse or death from any cause.
For AML and in Phase II only: Complete Remission (CR) Rate | From the date of first response up to end of study (approximately 1.5 years)
  Defined as the number of patients who achieve a CR as Best Response, divided by the number of participants in the analysis population.
For AML and in Phase II only: Complete Remission and Complete Remission with Partial Hematologic Recovery (CR/CRh) Rate | From the date of first response up to end of study (approximately 1.5 years)
  Defined as the number of patients who achieve a CR or CRh or CRi as best response, divided by the number of participants in the analysis population.
For AML and in Phase II only: Overall Response Rate (ORR: CRc + CRh + MLFS + PR) | From the date of first response up to end of study (approximately 1.5 years)
  Defined as the number of participants who achieve CR, CRi, CRh, MLFS or PR as best response, divided by the number of participants in the analysis population.
Rate of conversion from transfusion-dependence to transfusion-independence | From the date of first response up to end of study (approximately 1.5 years)
  Defined as the proportion of participants being post-baseline transfusion independent from baseline transfusion dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — ASST Papa Giovanni XXIII
Locations (11):
- France (4):
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hotel-Dieu, Nantes
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Italy (6):
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Hospital Universitari i Politècnic La Fe, Valencia, Spain